CLINICAL TRIAL: NCT06176781
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase III Clinical Trial to Evaluate the Efficacy and Safety of Edaravone Dexborneol Sequential Therapy in the Treatment of Patients With Acute Ischemic Stroke
Brief Title: The Efficacy and Safety of Edaravone Dexborneol Sequential Therapy in the Treatment of Patients With AIS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Simcere Pharmaceutical Co., Ltd (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SIM0308-302
Record Dates: First submitted 2023-12-11; First posted 2023-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Subjects With Acute Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequential group (Experimental): Edaravone Dexborneol concentrated solution for injections 37.5 mg BID administered intravenously for 5 - 10 days, and then followed by Edaravone Dexborneol Sublingual Tablets 30 mg BID administered sublingually for the last days, the total duration of treatment was 14 days
  Interventions: Drug: Edaravone Dexborneol Sequential Therapy
- Placebo group (Placebo Comparator): Injection Simulants(Edaravone Dexborneol concentrated solution for injections) administered intravenously for 5 - 10 days, and then followed by Sublingual Tablet Simulants(Edaravone Dexborneol Sublingual Tablets) BID administered sublingually for the last days, the total duration of treatment was 14 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Edaravone Dexborneol Sequential Therapy — Sequential treatment started with intravenous injection of edaravone dextrocamphorol 37.5 mg, twice a day for 5-10 days. Then, Edaravone Dexborneol Sublingual Tablets 36.0 mg was taken sublingual twice a day for 14 days (the total course of the two drugs was 14 days, a total of 28 times).
  Arms: Sequential group
Drug: Placebo — Injection Simulants(Edaravone Dexborneol concentrated solution for injections) administered intravenously for 5 - 10 days, and then followed by Sublingual Tablet Simulants(Edaravone Dexborneol Sublingual Tablets) BID administered sublingually for the last days, the total duration of treatment was 14 days
  Arms: Placebo group

SUMMARY:
SIM0308-302 is a multicenter, randomized, double-blind, placebo-controlled clinical III trial with the primary objective of evaluating the efficacy of Edaravone Dexborneol sequential therapy, consisting of Edaravone Dexborneol Injections followed by Edaravone Dexborneol Sublingual Tablets for total 14 days, in patients with acute ischemic stroke (AIS). The subject has a clinical diagnosis of AIS, within 48 hours from stroke onset to start of study treatment, with a National Institutes of Health Stroke Scale (NIHSS) between 6 and 20, had a total score of upper and lower limbs on motor deficits ≥ 2. The primary outcome is the proportion of subjects with modified Rankin scale score ≤ 2 at 90 days after treatment.

DETAILED DESCRIPTION:
SIM0308-302 is a multicenter, randomized, double-blind, placebo-controlled clinical III trial with the primary objective of evaluating the efficacy of Edaravone Dexborneol sequential therapy, consisting of Edaravone Dexborneol Injections followed by Edaravone Dexborneol Sublingual Tablets for total 14 days, in patients with acute ischemic stroke (AIS). The subject has a clinical diagnosis of AIS, within 48 hours from stroke onset to start of study treatment, with a NIHSS score between 6 and 20, had a total score of upper and lower limbs on motor deficits ≥ 2. The primary outcome is the proportion of subjects with modified Rankin scale score ≤ 1 at 90 days after treatment. The secondary outcomes included mRS score on day 90, the proportion of subjects with mRS score ≤2 on day 90, the change of NIHSS score from baseline to day 14 and the proportion of subjects with NIHSS score ≤1 on day 14, 30, 90 after treatment. Safety outcomes included adverse events, treatment related adverse events within day 90, and changes in vital signs and laboratory data before and after treatment.

Subjects in the Sequential group receive Edaravone Dexborneol concentrated solution for injections 37.5 mg BID administered intravenously for 5 - 10 days, and then followed by Edaravone Dexborneol Sublingual Tablets 30 mg BID administered sublingually for the last days, the total duration of treatment was 14 days. Subjects in the Placebo group receive placebo for 14 days. All the subjects were followed up to day 90 after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* 1. Aged from 18 to 80 years old, male or female; 2. Baseline National Institutes of Health Stroke Scale (NIHSS) score between 6 and 20, a sum scores of the fifth upper limb and the sixth lower limb ≥2 at admission; 3. AIS symptom onset within 48 hours, onset time defined as when the patient was last known to be well; 4. According to the "Diagnostic criteria of cerebrovascular diseases in China (version 2019)", patients were diagnosed with ischemic stroke, with their first onset or recovered well after the last onset (mRS score ≤ 1 point before this onset); 5. Informed consent from the patient or legally authorized representative.

Exclusion Criteria:

* 1. Intracranial bleeding disorders which were confirmed by cranial computed tomography scan, including hemorrhagic stroke, epidural hematoma, intracranial hematoma, intraventricular hemorrhage, subarachnoid hemorrhage, etc; 2. Severe disturbance of consciousness: NIHSS category 1a for consciousness >1; 3. Transient ischemic attack (TIA); 4. Systolic blood pressure ≥ 220 mmHg or diastolic blood pressure ≥ 120 mmHg after blood pressure control; 5. Severe mental disorder and dementia; 6. Alanine aminotransferase or aspartate transaminase > 2.0 × upper limit of normal value (ULN) or with known liver disorder, such as acute hepatitis, chronic active hepatitis, hepatic cirrhosis, etc； 7. Known kidney disease, renal insufficiency, serum creatinine > 1.5 × ULN or creatinine clearance < 50mL/min； 8. Received neuroprotective agents after this onset, including commercially available edaravone, edaravone dexborneol injection，nimodipine, ganglioside, citicoline, piracetam, butylphthalide, urinary kallidinogenase, etc； 9. Received or planed Embolectomy or interventional therapy after this onset； 10. Concurrent malignant tumor or currently receive antitumor treatment； 11. Severe systemic disease and life expectancy < 90 days; 12. Allergies to edaravone, dexborneol, or the excipients; 13. Pregnant or lactating patients or patients who plan to become pregnant; 14. History of a major surgery within 4 weeks before enrollment; 15. Participated in other clinical trials within 30 days before randomization or currently involved in other clinical trials; 16. Investigators consider they are not suitable for this trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 880 (Estimated)
Dates: Start 2023-12-28 (Estimated); Primary Completion 2025-03-28 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects with modified Rankin scale score ≤ 1 on 90 days after treatment | on 90 days
  To evaluate whether the proportion of subjects with mRS≤1 on the 90th day after treatment in the two groups meet the expected hypothesis

IPD SHARING:
Plan to Share IPD: No